CLINICAL TRIAL: NCT00034268
Title: A Phase 3 Trial of LY900003 Plus Gemcitabine and Cisplatin Versus Gemcitabine and Cisplatin in Patients With Advanced, Previously Untreated Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6428; H7X-MC-JVAA
Record Dates: First submitted 2002-04-24; First posted 2002-04-25 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: non-small cell lung cancer; Stage IIIB or IV non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ISIS 3521

INTERVENTIONS:
Drug: LY900003

SUMMARY:
The purposes of this study are to determine:

1. If treatment with LY900003 plus gemcitabine and cisplatin can help you live longer, compared with gemcitabine and cisplatin alone.
2. The safety of LY900003 plus gemcitabine and cisplatin and any side effects that might be associated with the combination of these three drugs.
3. Whether LY900003 plus gemcitabine and cisplatin can make your tumor smaller or disappear, and for how long, compared with gemcitabine and cisplatin alone.

It is possible that information collected during this study will be analyzed by the sponsor in the future to evaluate LY900003 plus gemcitabine and cisplatin for other possible uses or for other medical or scientific purposes other than those currently proposed.

LY900003 may not add any benefit to gemcitabine plus cisplatin.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IIIB or IV non-small lung cancer
2. Able to visit the doctor's office
3. At least 18 years of age
4. Adequate kidney, adrenal, and liver function

Exclusion Criteria:

1. Prior chemotherapy or biologic therapy for NSCLC
2. Central nervous system tumors
3. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03

CONTACTS AND LOCATIONS:
Locations (105):
- United States (20):
  - Hot Springs, Arkansas
  - Springdale, Arkansas
  - Los Angeles, California
  - Santa Rosa, California
  - Denver, Colorado
  - Fort Collins, Colorado
  - Wilmington, Delaware
  - Tucker, Georgia
  - Indianapolis, Indiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Robbinsdale, Minnesota
  - Latham, New York
  - New York, New York
  - Arlington, Texas
  - Dallas, Texas
  - Abingdon, Virginia
  - Marshfield, Wisconsin
- Argentina (2):
  - Mendoza, Mendoza Province
  - Ciudad de Buenos Aires
- Belgium (5):
  - Brasschaat
  - Edegem
  - Liège
  - Merksem
  - Ostend
- Las Condes, Santiago Metropolitan, Chile
- France (8):
  - Brest
  - Nice
  - Paris
  - Pessac
  - Rouen
  - Saint-Herblain
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (14):
  - Frankfurt am Main, Hesse
  - Augsburg
  - Berlin
  - Freiburg im Breisgau
  - Grobhansdorf
  - Hamburg
  - Heidelberg
  - Hofheim
  - Koin
  - Leipzig
  - München
  - Neustadt/Suedharz
  - Trier
  - Ulm
- Budapest, Hungary
- India (5):
  - Bangalore, Karnataka
  - Mumbai, Maharashtra
  - Pune, Maharashtra
  - Ludhiana, Punjab
  - New Dehli
- Italy (5):
  - Rozzano, Milano
  - Perugia
  - Pisa
  - Ravenna
  - Roma
- Netherlands (6):
  - 's-Hertogenbosch
  - Amsterdam
  - Arnhem
  - Groningen
  - Nieuwegien
  - Zwolle
- Oslo, Norway
- Poland (4):
  - Otwock, Masovian Voivodeship
  - Warsaw, Warszawa
  - Krakow-Nowa Huta
  - Wroclaw
- Puerto Rico (2):
  - Bayamón
  - Ponce
- Cluj-Napoca, Cluj, Romania
- Moscow, Russia
- South Africa (5):
  - Overport, Durban
  - Arcadia, Gauteng
  - Durban
  - Parklands
  - Tygerberg
- Spain (10):
  - Alicante, Alicante
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Madrid, Madrid
  - Palma de Mallorca, Palma de Mallorca
  - Oviedo, Principality of Asturias
  - Valencia, Valenica
  - Barakaldo, Vizcaya
  - Zaragoza, Zaragoza
- Sweden (3):
  - Linköping
  - Lund
  - Stockhlom
- Zurich, Switzerland
- Taiwan (3):
  - Taoyuan District, Kuei-Shan
  - Taichung, Taiwan, Province of China
  - Taipei
- United Kingdom (7):
  - Hull, East Yorkshire
  - London, Greater London
  - Southampton, Hampshire
  - Nottingham, Nottinghamshire
  - Glasgow, Scotland
  - Cardiff, South Glamorgan
  - Newcastle upon Tyne, Tyneside